CLINICAL TRIAL: NCT03434470
Title: Liver Elastography in Patients Undergoing Treatment for Hepatitis C - a Longitudinal Study
Brief Title: Liver Elastography in Patients Undergoing Treatment for Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1902
Record Dates: First submitted 2018-01-24; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Hepatitis C Virus Infection
Keywords: Ultrasound; Shear wave elastography; SWE; Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
According to the guidelines for treating hepatitis C livers stiffness (LS) measurement is equivalent to liver biopsy to prove grade-2 fibrosis or more by Metavir-score. Also flares of inflammation in other viral hepatitis (B) have been reported to increase the elastography measurements. There are very few reports so far on longitudinal data in a treatment cohort. In this study investigators will follow patients who undergo active treatment for hepatitis C virus (HCV). Investigators will collect longitudinal data of liver elastography and compare this to the current status of liver inflammation by blood samples. This may be important in order to know if transcutaneous US with elastography can be used as a tool to monitor active inflammation in liver disease and to quantify how much the inflammatory component contribute to LS and finally if it is possible to reverse not only inflammation but also liver fibrosis by treating viral hepatitis. Our aim is to assess shear wave elastography (SWE) and investigate if the method can be used, not only to define the indication for treatment through LS measurements, but also if LS due to inflammation and fibrosis may be reversible in treated patients. To investigate what role frequency of measurement obtains in follow up of patients with HCV play.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCV
* HCV RNA positive
* Approved for HCV treatment

Exclusion Criteria:

* Excessive alcohol use
* Pregnancy
* information of other cause of chronic liver disease (autoimmune hepatitis (AIH), primary sclerosing cholangitis (PSC), primary biliary cholangitis (PBC), Alpha-1-antitrypsin deficiency).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be HCV patients (n= 50), who will be invited to join the study consecutively as they have indication to start medical antiviral treatment for 8-, 12-, or 16 week, according to the genotype (1,2,3,4) and fibrosis stage.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Elastography | Baseline
  Obtained liver stiffness measurements (kPa) at baseline of participants receiving antiviral treatment.
Patient record | Baseline
  weight and height will be combined to report BMI in kg/m^2 at baseline of participants receiving antiviral treatment.
Biochemical analyses | Baseline
  Transaminases; aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT). Marker panels of liver fibrosis including AST to Platelet Ratio Index (APRI) and Fibrosis-4 index (FIB-4)will be calculated, at baseline of participants receiving antiviral treatment.
B-mode evaluation of the liver | Baseline
  Evaluation of Liver angle (acute/blunt), Steatosis (yes/no), Liver capsule (regular/irregular), Liver parenchyma (normal/coarse) at baseline of participants receiving antiviral treatment.

SECONDARY OUTCOMES:
Elastography | 3 months
  Obtained liver stiffness measurements (kPa) after end treatment (EOT).
Elastography | 6 months
  Obtained liver stiffness measurements (kPa), 3 months after end of treatment (EOT).
Elastography | 12 months
  Obtained liver stiffness measurements (kPa), 1 year after EOT.
B-mode evaluation of the liver | 3 months
  Evaluation of Liver angle (acute/blunt), Steatosis (yes/no), Liver capsule (regular/irregular), Liver parenchyma (normal/coarse) at at end of treatment (EOT).
B-mode evaluation of the liver | 6 months
  Evaluation of Liver angle (acute/blunt), Steatosis (yes/no), Liver capsule (regular/irregular), Liver parenchyma (normal/coarse), 3 months after end treatment (EOT).
B-mode evaluation of the liver | 12 months
  Evaluation of Liver angle (acute/blunt), Steatosis (yes/no), Liver capsule (regular/irregular), Liver parenchyma (normal/coarse), 1 year after EOT.
Patient record | 3 months
  weight and height will be combined to report BMI in kg/m^2 at end of treatment (EOT).
Patient record | 6 months
  weight and height will be combined to report BMI in kg/m^2, 3 months after end treatment (EOT).
Patient record | 12 months
  weight and height will be combined to report BMI in kg/m^2, 1 year after EOT.
Biochemical analyses | 3 months
  Transaminases; aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT). Marker panels of liver fibrosis including APRI and FIB-4 index will be calculated, at end of treatment (EOT).
Biochemical analyses | 6 months
  Transaminases; aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT). Marker panels of liver fibrosis including APRI and FIB-4 index will be calculated, 3 months after EOT.
Biochemical analyses | 12 months
  Transaminases; aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT). Marker panels of liver fibrosis including APRI and FIB-4 index will be calculated, 1 year after EOT.

CONTACTS AND LOCATIONS:
Overall Officials: Anesa Mulabecirovic, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trelsgard AM, Mulabecirovic A, Leiva RA, Nordaas IK, Mjelle AB, Gilja OH, Havre RF. Multiparametric liver assessment in patients successfully treated for hepatitis C: a 4-year follow-up. Scand J Gastroenterol. 2024 Oct;59(10):1184-1191. doi: 10.1080/00365521.2024.2388691. Epub 2024 Sep 1. PMID 39219192